CLINICAL TRIAL: NCT00225355
Title: Insulin Sensitisation as a Novel Mechanism to Lessen Ischaemic Burden in Overweight Non-Diabetic Patients With Chronic Stable Angina: A Pilot Study
Brief Title: Rosiglitazone Versus Placebo in Chronic Stable Angina
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: British Heart Foundation (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GlasUniRosiPlacebo; Eudract no. 2004-000949-38
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Angina Pectoris; Metabolic Syndrome X
Keywords: Angina pectoris; Metabolic syndrome; Ischaemic heart disease
MeSH Terms: conditions — Angina Pectoris; Metabolic Syndrome; Coronary Artery Disease | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
We wish to see if the drug rosiglitazone, currently used in the treatment of type 2 diabetes, could be used as a new treatment for angina when compared with placebo in overweight subjects who do not have overt diabetes. The drug will be given for 3 months and the subjects will be have their angina tested, by way of exercise testing, angina quality of life questionnaire and 24-hour ECG monitoring before and after using the drug.

DETAILED DESCRIPTION:
Chronic stable angina is a common manifestation of ischaemic heart disease. Current mechanical therapies (percutaneous coronary intervention and coronary artery bypass grafting) and pharmacological therapies (nitrates, calcium channel blockers, betablockers and potassium channel activators) main actions are to treat the end product of ischaemic heart disease on chronic stable angina, i.e. the flow limiting stenosis. We postulate that by treating insulin resistance, an upstream factor in the pathogenesis of ischaemic heart disease, we will improve angina by in turn improving endothelial function. We will attempt to demonstrate this by way of full bruce protocol exercise tolerance test, Seattle Angina Questionnaire and 24 hour ST segment analysis before and after treatment with the insulin sensitiser rosiglitazone for three months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable angina - to see if this improves
* Previous positive exercise tolerance test - to ensure that repeating it yields a result
* Disease not suitable for coronary intervention (Coronary artery bypass grafting or angioplasty) - so that best routine care is not withheld
* Do not have overt diabetes - work on this is being undertaken elsewhere
* Body mass index (BMI) greater than 25

Exclusion Criteria:

* Diabetes mellitus - see above
* Liver failure (ALT>70U/l, AST>80U/l)
* Renal failure (creatinine > 130mmol/l)
* Cardiac failure - rosiglitazone is contraindicated in those with NYHA 3 and 4 cardiac failure
* Physical disability - if it precludes treadmill testing
* Women of child bearing capacity
* Breast feeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-02; Study Completion 2006-11 (Estimated)

PRIMARY OUTCOMES:
Change in angina status at three months

SECONDARY OUTCOMES:
Change in pulse wave velocity at three months
Change in small vessel function at three months
Change in markers of haemostasis at three months
Change in biochemical markers of insulin resistance/metabolic syndrome at three months
Change in blood pressure at three months
Change in anthropometric status at three months

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, MBChB PhD, Principal Investigator — University of Glasgow; Stuart M Cobbe, MBChB MD, Principal Investigator — University of Glasgow
Locations (1):
- Cardiology Department, Glasgow Royal Infirmary, Glasgow, United Kingdom